CLINICAL TRIAL: NCT02713061
Title: An Open-label Phase 2 Study to Evaluate the Safety and Immnogenicity of a Single Subcutaneous Injection of Quadrivalent TAK-850 in Healthy Adult Subjects
Brief Title: A Phase 2 Study of a Subcutaneous Injection of TAK-850 in Healthy Adult Participants
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-850/CPH-004; U1111-1178-8045 (Registry Identifier: WHO)
Record Dates: First submitted 2016-03-15; First posted 2016-03-18 (Estimated); Last update posted 2016-08-25 (Estimated); Status verified 2016-08

CONDITIONS: Influenza Prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TAK-850 0.5 mL (Experimental): TAK-850 0.5 mL (15 µg of hemagglutinin [HA] antigen per strain), subcutaneous injection, once on Day 1.
  Interventions: Drug: TAK-850

INTERVENTIONS:
Drug: TAK-850 — TAK-850 injection

SUMMARY:
This clinical trial is a Phase 2 study of a single subcutaneous injection of TAK-850 for 22 days in healthy Japanese adults.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the safety and immunogenicity of a single subcutaneous injection of TAK-850 for 22 days in healthy Japanese adults.

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator, the participant is capable of understanding and complying with protocol requirements.
2. The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.
3. The participant is a healthy Japanese adult male or female.
4. The participant is aged 20 to 49 years, inclusive, at the time of informed consent.
5. The participant has a body mass index (BMI) between 18.5 and 25.0 kg/m^2, inclusive, at the time of eligibility evaluation.
6. If the participant is a female of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent throughout the duration of the study.

Exclusion Criteria:

1. The participant has received any investigational compound within 4 months prior to the initial injection of study vaccine.
2. The participant has been vaccinated with seasonal influenza vaccine within 6 months prior to the initial injection of study vaccine.
3. The participant has a history of influenza infection within 6 months prior to the initial injection of study vaccine
4. The participant has been vaccinated with TAK-850 (trivalent).
5. The participant is a study site employee, an immediate family member of such an employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling), or may consent under duress.
6. The participant has uncontrolled, clinically significant manifestations of neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, endocrine or other disorders, which may impact the ability of the participant to participate or potentially confound the study results.
7. The participant has an oral temperature ≥37.5°C prior to the initial injection of study vaccine on Day 1.
8. The participant has any medically diagnosed or suspected immune deficient condition.
9. The participant has an immune compromising condition or disease, or is currently undergoing a form of treatment or was undergoing a form of treatment that can be expected to influence immune response within 30 days prior to the initial injection of study vaccine. Such treatments include, but is not limited to, systemic or high dose inhaled corticosteroids (>800 μg/day of beclomethasone dipropionate or equivalent; the use of inhaled and nasal steroids that do not exceed this level will be permitted), radiation treatment or other immunosuppressive or cytotoxic drugs.
10. The participant has received antipyretics within 4 hours prior to the initial injection of study vaccine.
11. The participant has a history of Guillain- Barré Syndrome, demyelinating disorders (including acute disseminated encephalomyelitis [ADEM] and multiple sclerosis) or convulsions.
12. The participant has a functional or surgical asplenia.
13. The participant has a rash, other dermatologic conditions or tattoos which may interfere with the evaluation of injection site reaction as determined by the Investigator.
14. The participant has a history of, or is infected with the Hepatitis B Virus (HBsAgs), Hepatitis C Virus (HCV) or Human Immunodeficiency Virus (HIV).
15. The participant has a known hypersensitivity to any component of TAK-850.
16. The participant has a history of severe allergic reactions or anaphylaxis.
17. The participant has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 1 year prior to the initial injection of study vaccine or is unwilling to agree to abstain from alcohol and drugs throughout the study.
18. The participant has received any blood products (e.g. blood transfusion or immunoglobulin) within 90 days prior to the initial injection of study vaccine.
19. The participant has received a live vaccine within 4 weeks (28 days) or an inactivated vaccine within 2 weeks (14 days) prior to the initial injection of study vaccine.
20. If female, the participant is pregnant or lactating or intending to become pregnant before signing informed consent, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
21. The participant has donated whole blood ≥200 mL within 4 weeks (28 days), ≥400 mL within 12 weeks (84 days), ≥800 mL within 52 weeks (364 days), or blood components within 2 weeks (14 days) prior to the initial injection of study vaccine.
22. The participant has abnormal laboratory values that suggest a clinically significant underlying disease at the assessment prior to the initial injection of study vaccine, or the participant has the following lab abnormalities: alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) more than 3 times the upper limits of normal.
23. In the opinion of the investigator or sub-investigator, the participant is unlikely to comply with protocol requirements or is considered ineligible for any other reason.

Ages: 20 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Up to Day 22
  An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment The adverse events will include solicited local and systemic AEs.
Seroprotection Rate of Hemagglutination Inhibition (HI) Antibody Titer (egg-derived antigen) | Day 22
  Seroprotection Rate is defined as the percentage of participants with HI antibody titer ≥ 40 for each of the four strains (A/H1N1 strain, A/H3N2 strain, B/Yamagata strain, B/Victoria strain).
Seroconversion Rate of HI Antibody Titer (egg-derived antigen) | Day 22
  Seroconversion Rate is defined as the percentage of participants with a baseline HI antibody titer of ≥ 10 achieving a minimal 4-fold increase, or baseline HI antibody titer of < 10 achieving an HI antibody titer of ≥ 40 for each of the four strains (A/H1N1 strain, A/H3N2 strain, B/Yamagata strain, B/Victoria strain).
Geometric Mean Fold Increase (GMFI) in HI Antibody Titer (egg-derived antigen) | Day 22

SECONDARY OUTCOMES:
Number of Participants who Meet the Markedly Abnormal Criteria for Vital Sign Measurements | Day 22
  Vital signs will include blood pressure, pulse rate and respiratory rate.
Number of Participants who Meet the Markedly Abnormal Criteria for Safety Laboratory Tests | Day 22
  Laboratory tests will include hematology, biochemistry and urinalysis tests.
Geometric Mean Titer (GMT) of HI Antibody Titer (egg-derived antigen) | Day 22
Seroprotection Rate of Single Radial Hemolysis (SRH) Antibody Titer (egg-derived antigen) | Day 22
  Seroprotection Rate is defined as the percentage of participants with SRH antibody titer ≥ 25 mm^2 for each of the four strains (A/H1N1 strain, A/H3N2 strain, B/Yamagata strain, B/Victoria strain).
Seroconversion Rate of SRH Antibody Titer (egg-derived antigen) | Day 22
  Seroconversion Rate is defined as the percentage of participants with a baseline SRH antibody titer of ≥ 4 mm^2 achieving a minimal 50 percent increase, or baseline HI antibody titer of < 4 mm^2 achieving an SRH antibody titer of ≥ 25 mm^2 for each of the four strains (A/H1N1 strain, A/H3N2 strain, B/Yamagata strain, B/Victoria strain).
GMFI in SRH Antibody Titer (egg-derived antigen) | Day 22
GMT of SRH Antibody Titer (egg-derived antigen) | Day 22
Seroprotection Rate of HI Antibody Titer (cell-derived antigen) | Day 22
  Seroprotection Rate is defined as the percentage of participants with HI antibody titer ≥ 40 for each of the four strains (A/H1N1 strain, A/H3N2 strain, B/Yamagata strain, B/Victoria strain).
Seroconversion Rate of HI Antibody Titer (cell-derived antigen) | Day 22
  Seroconversion Rate is defined as the percentage of participants with a baseline HI antibody titer of ≥ 10 achieving a minimal 4-fold increase, or baseline HI antibody titer of < 10 achieving an HI antibody titer of ≥ 40 for each of the four strains (A/H1N1 strain, A/H3N2 strain, B/Yamagata strain, B/Victoria strain).
GMFI in HI Antibody Titer (cell-derived antigen) | Day 22
GMT of HI Antibody Titer (cell-derived antigen) | Day 22
  GMT of HI antibody titer for each of the four strains (A/H1N1 strain, A/H3N2 strain, B/Yamagata strain, B/Victoria strain), 21 days after vaccination.
Seroprotection Rate of SRH Antibody Titer (cell-derived antigen) | Day 22
  Seroprotection Rate is defined as the percentage of participants with SRH antibody titer ≥ 25 mm^2 for each of the four strains (A/H1N1 strain, A/H3N2 strain, B/Yamagata strain, B/Victoria strain).
Seroconversion Rate of SRH Antibody Titer (cell-derived antigen) | Day 22
  Seroconversion Rate is defined as the percentage of participants with a baseline SRH antibody titer of ≥ 4 mm^2 achieving a minimal 50 percent increase, or baseline HI antibody titer of < 4 mm^2 achieving an SRH antibody titer of ≥ 25 mm^2 for each of the four strains (A/H1N1 strain, A/H3N2 strain, B/Yamagata strain, B/Victoria strain).
GMFI in SRH Antibody Titer (cell-derived antigen) | Day 22
GMT of SRH Antibody Titer (cell-derived antigen) | Day 22

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Toshima-ku, Tokyo, Japan